CLINICAL TRIAL: NCT01003613
Title: Evaluation of Tranilast as Adjunctive Therapy Before Primary Pterygium Excision Compared With Conjunctival Autograft
Brief Title: Evaluation of Tranilast to Treat Pterygium Before Excision
Acronym: TPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gildasio Castello de Almeida Junior (Other)
Collaborators: Hospital de Base (Other)
Responsible Party: Sponsor-Investigator, Gildasio Castello de Almeida Junior, Prof. Dr., FAMERP, Sao Jose do Rio Preto Medical School
Organization: Sao Jose do Rio Preto Medical School (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3049/2009
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-03

CONDITIONS: Pterygium
Keywords: Tranilast; fibrin glue; primary pterygium; conjunctival autograft
MeSH Terms: conditions — Pterygium | interventions — tranilast; Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranilast (Active Comparator): CAT with FG and Tranilast and MMC 0.02%
  Interventions: Drug: Tranilast, and Tissucol
- Control (Placebo Comparator): CAT with FG and MMC 0.02%
  Interventions: Other: Beriplast P

INTERVENTIONS:
Drug: Tranilast, and Tissucol — 1.0%, 0.1 ml, subconjunctival route, single dose
  Other Names: Rizaben, Tissucol
  Arms: Tranilast
Other: Beriplast P — 0.1 ml to attach graft
  Other Names: Tissucol
  Arms: Control

SUMMARY:
Recurrent or secondary pterygium often has often a growing fibrovascular tissue more exuberant than the primary. Histological findings differ from the primary, since the typical changes in the degenerate connective tissue are absent. The strong immunoreactivity and release of basic fibroblast growth (b-FGF) in cultured fibroblasts of recurrent pterygia suggest that fibroblasts may play an important role in pterygium recurrence. Tranilast used is an antiallergic drug that has an inhibitory effect on the release of chemical transmitters, such as histamine and leukotrienes from mast cells as well as a suppressive effect on vascular permeability.This drug also reduces TGF-β1 production and collagen synthesis in various cells. Tranilast might reduce pterygium recurrence by suppressing TGF-β1 synthesis in conjunctival fibroblast after pterygium surgery. The investigators want to confirm these findings and also compare the recurrence rate between the two types of surgery. Tranilast might be an alternative of mitomycin use, and also less toxic. This study aim to compare the effectiveness of preventing recurrence by using tranilast by topical subconjunctival administration previous to conjunctival autograft transplantation surgery in cases of primary pterygium, and will be perform clinical evaluation and TGF-beta-1 immunohistochemical detection by the anti-TGF-beta 1 antibody as well as fibroblast culture.

DETAILED DESCRIPTION:
This is a prospective, randomised, control trial of 50 participants. Twenty five patients in each arm. Twenty five patients undergo standard pterygium excision with the fibrin glue (Tissucol) conjunctival autograft . Twenty five patients undergo pterygium surgery with fibrin glue (Tissucol), and subconjunctival injection of 0.1 ml of Tranilast 1.0% in the head of pterygium 30 days before surgery. Participants will be reviewed, selected, and consented on a pre-assessment day. Surgery will be performed 4 at a time on an all day surgery operating list. Randomisation of the surgery type will be done at the time of surgery after the pterygium has been excised and the autograft taken. The surgeries will perform by a single surgeon (Almeida Jr, GC). Follow-up will occur at week 1,4, 26, 52. Slit lamp examination will indicate pterygium recurrence. Corneal recurrence will consider when it 0.5 mm of invaded conjunctival tissue,in the clear cornea from the anatomical limbus. The conjunctival recurrence will consider of any size conjunctive fibrovascular invasion inside the graft. The localization and of immunohistochemical will be perform for TGF-B.

ELIGIBILITY:
Inclusion Criteria:

* Primary pterygium

Exclusion Criteria:

* Keratoconjunctivitis sicca
* Sjögren disease
* Vernal keratoconjunctivitis
* Acne rosacea
* Neurotrophic keratopathy
* Severe dysfunction of the meibomius glands
* Use of any immunosuppressive drug, through systemic and topical route
* Aged under 18 years of age and vulnerable groups
* Glaucoma and use of ocular hipotensor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Recurrence rate at months six and twelve months Immunohistochemical and cell morphology analysis at the end of study, 12 months | 6 and 12 months

SECONDARY OUTCOMES:
Patient discomfort at day one, six and twelve months Safety of Tranilast | one day, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gildasio C Almeida Jr, Prof Dr, Principal Investigator — Sao Jose do Rio Preto Medical School; Sidney JF Sousa, Prof Dr, Study Chair — USP - Ribeirão Preto; Reinaldo Azoubel, Prof Dr, Study Director — Prof Dr; Vinicius Tadeu NS Nascimento, Student, Study Chair — Sao Jose do Rio Preto Medical School; Acacio AS Lima Filho, MD, Study Chair — Federal University of São Paulo
Locations (1):
- Hospital de Base/FAMERP, São José do Rio Preto, São Paulo, Brazil

REFERENCES:
- [Result] Wang M, Zhang JJ, Jackson TL, Sun X, Wu W, Marshall J. Safety and efficacy of intracapsular tranilast microspheres in experimental posterior capsule opacification. J Cataract Refract Surg. 2007 Dec;33(12):2122-8. doi: 10.1016/j.jcrs.2007.07.041. PMID 18053915
- [Result] Ji CN, Hu YZ, Ding ZP, Li GG. [The investigation of tranilast on the proliferation and migration of human Tenon's capsule fibroblasts]. Zhonghua Yan Ke Za Zhi. 2004 Mar;40(3):165-9. Chinese. PMID 15307986
- [Result] Yasukawa T, Kimura H, Dong J, Tabata Y, Miyamoto H, Honda Y, Ogura Y. Effect of tranilast on proliferation, collagen gel contraction, and transforming growth factor beta secretion of retinal pigment epithelial cells and fibroblasts. Ophthalmic Res. 2002 Jul-Aug;34(4):206-12. doi: 10.1159/000063884. PMID 12297693
- [Derived] Almeida Junior GC, Arakawa L, Santi Neto Dd, Cury PM, Lima Filho AA, Sousa SJ, Alves MR, Azoubel R. Preoperative tranilast as adjunctive therapy to primary pterygium surgery with a 1-year follow-up. Arq Bras Oftalmol. 2015 Jan-Feb;78(1):1-5. doi: 10.5935/0004-2749.20150002. PMID 25714528